CLINICAL TRIAL: NCT04285372
Title: A Randomized, Prospective, Post-market, Multicenter Study to Evaluate the Potential Benefit of Side Branch Ballooning, in the Setting of Single Stenting With Systematic Proximal Optimization Technique, in the Treatment of Bifurcation Lesion
Brief Title: Keep bIfurcation Single Stenting Simple
Acronym: KISS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ceric Sàrl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KISS
Record Dates: First submitted 2020-02-21; First posted 2020-02-26 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Coronary Disease
Keywords: Coronary disease; Bifurcation lesion
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): No intervention on the side branch in the context of percutaneous coronary intervention for the treatment of bifurcation lesion
  Interventions: Procedure: No side branch protection/ballooning
- Control group (Active Comparator): Side branch protection: Ballooning or Kissing Balloon Technique, in the context of percutaneous coronary intervention for the treatment of bifurcation lesion
  Interventions: Procedure: Side branch protection/ballooning

INTERVENTIONS:
Procedure: Side branch protection/ballooning — Side branch protection in the context of percutaneous coronary intervention for the treatment of bifurcation lesion
  Arms: Control group
Procedure: No side branch protection/ballooning — No intervention on the side branch
  Arms: Test group

SUMMARY:
KISS study is an investigator-initiated, multi-centre, prospective, randomized (1:1), parallel, two-arm, non-inferiority trial aiming to compare two bifurcation PCI procedures for Side Branch protection

DETAILED DESCRIPTION:
In the treatment of bifurcation lesion, the role of side branch intervention for improving the safety of Percutaneous Coronary Intervention (PCI), when MB is treated according to the Murray law with a Proximal Optimization Technique (POT), remains unclear.

The KISS study will evaluate the non-inferiority of no side branch intervention versus side branch ballooning, in the setting of single stenting with systematic proximal optimization technique.

ELIGIBILITY:
Inclusion Criteria:

1. Coronary artery disease requiring revascularization that is amenable to percutaneous coronary intervention (PCI)
2. Any de novo Medina type bifurcation lesion with >70% lesion in the main vessel by visual assessment except Medina 0,0,1 if the planned strategy does not include a main branch stenting
3. Side branch diameter compatible with a PCI with stent implantation (≥ 2.25mm)
4. Side branch requiring a protection wire according to operator evaluation
5. Anatomy compatible with a proximal optimization technique
6. Post main branch treatment (stenting then POT): Absence of side branch occlusion Or low flow associated with ongoing ischemia (either chest pain or ST changes)
7. Male or female patient >18 years old

Exclusion Criteria:

1. Acute myocardial infarction with ongoing ST-elevation
2. Cardiogenic shock
3. Requirement for ongoing hemodialysis
4. Life-expectancy limited to <12 months due to co-morbid condition
5. Lesion involves the left main coronary artery
6. Lesion requiring a double stenting
7. Plan to treat >1 other coronary vessel at the time of the index procedure
8. Two lesions treated in the same session: unsuccessful PCI on the single non bifurcation lesion in a non-target vessel before the treatment of the target lesion.
9. Chronic total occlusion of any target vessel
10. Left ventricular ejection fraction <20%
11. Side branch TIMI Flow <3
12. Pre-dilatation of the Side Branch during the procedure prior to randomization
13. Known allergy to Aspirin
14. Known allergy to Clopidorel and Prasugrel and Ticagrelor
15. Known allergy to stent drug elutant
16. Known allergy to any other component of Onyx Resolute stent
17. Ongoing participation in another investigational device or drug study
18. Inability to provide informed consent
19. Patients under judicial protection, tutorship or curatorship
20. Pregnant and breast-feeding women or intention to become pregnant prior to completion of all follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Periprocedural Myocardial infarction | up to 48 hours post-procedure, up to 12 months
  Rate of peri-procedural Myocardial Infarction (MI) at discharge or 48 hours post-procedure whichever comes first as judged by clinical evaluation in association with day-1 troponin evaluation using the ARC-2 definition

SECONDARY OUTCOMES:
Technical success (1) | Intraoperative, up to 12 months
  Deployment of main branch (MB) stent with <20% residual stenosis and a patent side branch at end of procedure upon corelab analysis
Technical success (2) | Intraoperative, up to 12 months
  Total procedure time
Technical success (3) | up to 12 months
  Acute gain in main and side branches as measured with a dedicated quantitative coronary analysis (QCA) software
Technical success (4) | Intraoperative, up to 12 months
  Fluoroscopy time
Technical success (5) | Intraoperative, up to 12 months
  Total radiation dose (air kerma)
Technical success (6) | Intraoperative, up to 12 months
  Total contrast dose
Technical success (6) | Intraoperative, up to 12 months
  Need to cross over (any intervention on SB in the test arm or failure to intervene on the SB in the control arm)
Target Lesion Failure (TLF) | 1 month and 12 months
  Composite of:
  * Cardiac Death
  * Target vessel Myocardial Infarction
  * Clinically driven Target lesion revascularization (ci-TLR)
Target Lesion Revascularization (TLR) | 1 month and 12 months
  Main Branch & Side Branch TLR
Stent thrombosis: | 1 month and 12 months
  Definite or Probable stent thrombosis (ARC-2 criteria)
Angina status | 1 month and 12 months
  Angina status according to the Canadian Cardiovascular Society (CCS) classification (Grade 1 to 4)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard CHEVALIER, MD, Principal Investigator — ICPS - Institut Cardiovasculaire Paris Sud
Locations (20):
- France (9):
  - CHU Caen, Caen
  - Hôpital Privé Dijon Bourgogne, Dijon
  - CHU Timone Adultes, Marseille
  - Hôpital Privé Jacques Cartier ICPS, Massy
  - Clinique du Pont de chaume, Montauban
  - CHU Nîmes, Nîmes
  - Hôpital Privé Claude Galien ICPS, Quincy-sous-Sénart
  - Clinique Saint Hilaire, Rouen
  - CHU Toulouse Rangueuil, Toulouse
- Italy (3):
  - Universita' Cattolica del Sacro Cuore, Roma
  - Istituto Clinico Humanitas, Rozzano
  - IRCCS Policlinico San Donato, San Donato
- Hospital de Santa Cruz, Lisbon, Portugal
- Spain (4):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital de Cabuenes, Gijón
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- CHUV Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- United Kingdom (2):
  - Freeman Hospital Newcastle, Newcastle, Tyne and Wear
  - Royal Sussex County Hospital, Brighton

IPD SHARING:
Plan to Share IPD: No